CLINICAL TRIAL: NCT03376854
Title: Pilot Randomized Clinical Trial of Therapeutic Hypothermia Plus Neuromuscular Blockade vs. Standard of Care in COVID-19 Patients With Moderate to Severe ARDS - the Cooling to Help Injured Lungs (CHILL) Pilot Study
Brief Title: Pilot RCT of Therapeutic Hypothermia Plus Neuromuscular Blockade in COVID-19 Patients With ARDS
Acronym: CHILL-pilot
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Competition from other studies and initiation of a larger multi center trial
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Jeffrey Hasday, Professor of Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00078506
Record Dates: First submitted 2017-12-07; First posted 2017-12-19 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Respiratory Distress Syndrome, Adult; Sars-CoV2
Keywords: COVID-19, ARDS, targeted temperature management
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19 | interventions — Hypothermia, Induced; Neuromuscular Blocking Agents

STUDY DESIGN:
Intervention Model Description: Randomized (1:1) control (non-blinded) trial
Masking Description: Since it will be obvious to observers of the subjects whether they are in the treatment (TH+NMB) or control groups, the study is not masked but all treatments that determine outcome are protocolized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Hypothermia + Neuromuscular blockade (Experimental): Deep sedation and Neuromuscular blockade (NMB) and surface temperature management to maintain core temperature between 34 and 35°C for 48h, then rewarm to 36°C at 0.33°C per h and NMB discontinued when core temp reaches 35.5°C.
  Interventions: Device: Hypothermia; Drug: Neuromuscular Blocking Agents
- Standard of care (Active Comparator): Acetaminophen and surface temperature management to maintain core temperature between 37°C and 38°C. Rewarming to 37°C for hypothermia ≤36°C with continuous renal replacement therapy.
  Interventions: Device: Standard of Care

INTERVENTIONS:
Device: Hypothermia — Subjects will be cooled using either cooling blankets or gel-pad systems to maintain core temperature 34-35°C.
  Other Names: Targeted temperature Management
  Arms: Hypothermia + Neuromuscular blockade
Drug: Neuromuscular Blocking Agents — Subjects in the TH + NMB arm will be deeply sedated using agents at the discretion of the primary ICU team, then start continuous iv infusion of either cisatracurium, atracurium, or vecuronium titrated to 2 twitches on train of four monitoring and further titrated to ablate visible shivering.
  Other Names: Paralytics
  Arms: Hypothermia + Neuromuscular blockade
Device: Standard of Care — Subjects who are hypothermic (≤36°C) during CRRT will receive surface warming to restore core temperature to 37°C. Patients with core temperature >38°C will receive 650 mg acetaminophen and, if temperature remains >38°C, surface cooling will be initiated to return core temperature to 37-38°C.
  Other Names: Usual temperature management
  Arms: Standard of care

SUMMARY:
Acute Respiratory Distress Syndrome (ARDS) is a serious condition that occurs as a complication of medical and surgical diseases, has a mortality of ~40%, and has no known treatment other than optimization of support. Data from basic research, animal models, and retrospective studies, case series, and small prospective studies suggest that therapeutic hypothermia (TH) similar to that used for cardiac arrest may be lung protective in patients with ARDS; however, shivering is a major complication of TH, often requiring paralysis with neuromuscular blocking agents (NMBA) to control. Since the recently completed NHLBI PETAL ROSE trial showed that NMBA had no effect (good or bad) in patients with moderate to severe ARDS, the investigators sought to evaluate whether TH combined with NMBA is beneficial in patients with ARDS. The investigators are scheduled to begin enrolling in a Department of Defense-funded Phase IIb multicenter RCT of TH (core temperature 34-35°C) + NMBA for 48h vs. usual temperature management in patients with ARDS with time on ventilator as the primary outcome. Since COVID-19 is now the most common cause of ARDS, we are conducting a pilot study to examine the safety and feasibility of including patients with COVID-19-associated ARDS in our upcoming trial. In this pilot, we will randomize 20 patients with COVID-19 and ARDS to either TH+NMBA for 48h or usual temperature management. The primary outcome is achieving and maintaining the target temperature. Secondary outcomes include safety, physiologic measures, mortality, hospital and ICU length of stay, and serum biomarkers collected on days 0, 1, 2, 3, 4, and 7.

DETAILED DESCRIPTION:
Background:

Despite recent advances in supportive care for patients with acute respiratory distress syndrome (ARDS), mortality remains >40%. Fever worsens and hypothermia mitigates animal models of ALI and in small non-randomized in patients with ARDS. Since hypothermia reduces oxygen utilization as long as shivering is blocked, TH may reduce injury in part by allowing lower levels of assisted ventilation. TH likely exerts additional lung protective effects by directly modifying temperature-dependent cellular processes in endothelium, epithelium, and leukocytes. Neuromuscular blockade (NMB) is the ultimate treatment to block shivering and is frequently used in patients with ARDS to facilitate ventilator management. Since the recently completed NHLBI PETAL ROSE trial showed that NMB caused conferred neither benefit nor harm in patients with moderate to severe ARDS, the investigators have bundled TH with NMB to reduce shivering. An open-label study of 8 ARDS patients showed that studying TH + NMB in patients with moderate to severe ARDS was feasible. Moreover, the patients treated with TH +NMB had more 28-day ventilator-free days (VFDs), ICU-free days (ICU-FDs) and greater hospital survival (75% vs. 25%; p = 0.027) than historical controls with ARDS and NMB but without TH. Within the limits of historical comparisons, these results support further study of TH in ARDS. A Department of Defense-funded Phase IIb multicenter trial of TH+NMB in patients with moderate to severe ARDS will begin enrolling in Fall, 2020. Since COVID-19 has become the most common cause of ARDS, it is important to understand whether patients with COVID-19-associated ARDS can be included in the multicenter trial.

Focus of Study: We will conduct a single-site feasibility and safety RCT pilot of TH+NMB for 48h vs. usual temperature management in 20 patients with COVID-19-associated ARDS. We will also analyze efficacy markers to help decide whether the treatment duration (48h) to be used in the multicenter trial is appropriate for patients with COVID-19-associated ARDS. The results of this pilot help us decide whether to include patients with COVID-19-associated ARDS in our planned multicenter trial of TH+NMB in ARDS from all causes or to pursue a separate trial focused on patients with COVID-19-associated ARDS.

Primary and secondary objectives: The primary objective is to assess the safety and feasibility of the 48h TH+NMB treatment protocol. The secondary objective is to compare the TH+NMB and control arms for efficacy markers to be used in the multicenter trial.

Study design: The CHILL trial is a single center RCT.

Intervention: The study intervention is TH to core temperature 34°-35°C + NMB for 48h. Patients in the TH+NMB arm will receive deep sedation, continuous infusion of cisatracurium and mechanical ventilation for at least 48h. Decisions about transition to unassisted breathing, extubation, and transfer from ICU will be based on criteria in the CHILL study protocol.

TH+NMB: Once sedation and NMB are confirmed, TH to 34°-35°C will be initiated using surface cooling. Temperature will be measured from a central probe. Once target temperature is reached, TH will be maintained for 48h. Patients will then be rewarmed to 35.5°C by 0.3°C/h and the cooling devices removed. Post-TH fever suppression is not part of the CHILL protocol and will be performed at the discretion of the primary ICU team. TH+NMB will be aborted for persistent severe bradycardia, uncontrolled bleeding, and intractable arrhythmias.

Usual temperature management: Patients will receive light sedation (RASS 0 to -1). During the 54h post-randomization treatment period, acetaminophen will be given for core temperature >38°C and surface cooling will be initiated if core temperature remains >38°C within ≥45 minutes of receiving acetaminophen and adjusted to maintain core temperature ≤38°C. If core temperature ≤36°C, patients in this arm will receive surface warming to core temperature 37°C. Following the 54h treatment period, temperature will be managed at the discretion of the primary ICU team.

Concomitant Treatment: Since prone positioning independently improves survival in ARDS, starting and stopping rules for prone positioning have been protocolized.

Primary and Secondary Endpoints:

Primary endpoint: The low and high core temperatures in each 2-hour period will be recorded for each of the first four study days. The time required to reach the target temperature and the percent of readings within the target range in the TH+NMB arm will be determined.

Secondary endpoints:

Clinical: (a) 28-day VFDs. The 28-day VFDs will be calculated at day 28. (b) 28-day ICU-FDs:. The 28-day ICU-FDs will be calculated at day 28; (c) day 0, 1, 2, 3, 4, and 7 non-neurologic SOFA score; (d) Glasgow coma score at hospital discharge; (e) 60- and 90-day survival; (f) 60- and 90-day functional status. The Montreal Cognitive Assessment Tool (MOCA) will be administered at ICU and hospital discharge.

Physiologic: (a) day-3 and -7 driving pressure; (b) day-3 and day-7 oxygen saturation index (OSI).

Plasma Biomarker: Day 0, 1, 2, 3, 4, and 7 plasma IL-1ß, IL-6, IL-8, IL-18, soluble-RAGE, surfactant protein-D, soluble ICAM-1, MMP8, and soluble TNFRI.

Safety:

1. For the first 54h: (a) continuous cardiac monitoring for bradycardia with associated hypotension requiring i.v. fluid or vasopressors; (b) every 6h blood glucose measurement; (c) every 12 h potassium, magnesium and phosphate; (d) significant bleeding event (requiring 2u packed red blood cells or surgical or interventional radiologic intervention)
2. First 7 days: (a) Ventilator-associated pneumonia (VAP); (b) other secondary infections; (c) monitor for SAEs

Schedule of Clinical and Laboratory Evaluations:

1. Definitions:

   1. Day 0: day of randomization
   2. Comprehensive metabolic panel (CMP): includes basic electrolytes, BUN, creatinine, ALT, AST, alkaline phosphatase, bilirubin, calcium, magnesium, phosphate, C-reactive protein (CRP)
   3. CBC: complete blood count
   4. Driving Pressure = Plateau Pressure - PEEP with patient NOT making inspiratory effort (on NMB or post-NMB and observed RR at set ventilator rate)
   5. OSI = Mean airway pressure x 100 x FIO2/SpO2
2. Clinical and Research laboratory testing: Two purple top (EDTA; 14 ml blood) tubes will be collected for biomarker analysis at randomization and on study days 1, 2, 3, 4, and 7 at 8:00-10:00 on study days 1, 2, 3, 4, and 7. Clinical laboratory testing required for secondary clinical outcomes at enrollment and on study days 1, 2, 3, 4, and will be performed as part of usual clinical care whenever possible) at 6:00-10:00 AM and 6:00-10:00 PM
3. Day -2 to 0 (Screening and enrollment): To facilitate randomization within the inclusion window, we will consent and enroll based on partial fulfillment of randomization criteria and randomize once all criteria are met. Patients with COVID-19, receiving mechanical ventilation for ≤7 days and have bilateral pulmonary opacities not fully explained by pleural effusions, atelectasis, or hydrostatic pulmonary edema for <48h will be offered enrollment and will be randomized when P/F ratio is <200. In patients without arterial blood gas values, the P/F ratio will be inferred from SpO2 readings as described by Brown et al. (Chest 150:307; 2016).

   1. Pregnancy testing in women of child-bearing years
   2. Obtain informed consent from patient or Legally Authorized Representative (LAR) depending on capacity
   3. Complete Screening, enrollment, and randomization CRFs.
   4. If P/F<200 at enrollment, proceed with randomization, otherwise follow until P/F < 200 or patient exits the 48 hr ARDS or 7 day mechanical ventilation windows.

3. Day 0 (Randomization day): Pt. identified in screen:

1. Obtain baseline plasma for research testing. If >8h since last CBC and CMP or >24 since last CRP, send new samples to lab.
2. Randomize.
3. If patient does not have a central temperature probe, place esophageal probe.
4. For TH+NMB arm, confirm adequate sedation (RASS -4) and NMB (Train of four ≤2 twitch) and initiate TH protocol.
5. Complete Randomization Worksheet and Randomization and Baseline Data CRFs
6. Note time cooling initiated and time patient first reached target temperature on Baseline CRF

   4.Day 1-4:

a. Fill out Daily CRFs b. Collect plasma for research testing. c. Measure Driving Pressure and OSI d. Make sure CBC and CMP sent every 12h and CRP every 24h e. Rewarming starts after 48h cooling on day 3 f. Complete Unassisted Breathing Checklist form if applicable g. Assess for adverse events

5. Days 5-6:

a. Follow for ventilator status, ICU status, survival, SAEs b. Follow CRP daily c. Complete Unassisted Breathing Checklist form if applicable d. Assess for adverse events

6. Day 7:

a. Fill out Day 7 CRF b. Collect plasma for research testing. c. Measure Driving Pressure and OSI d. Make sure CBC, CMP, and CRP sent e. Complete Unassisted Breathing Checklist form if applicable f. Assess for adverse events

7. Day 8-27:

a. Follow for ventilator status, ICU status, survival, SAEs b. Complete Unassisted Breathing Checklist form if applicable

8. Day 28:

1. Complete Day 28 CRF
2. Calculate 28 day VFDs and ICU-FDs

   9. When patient is discharged from the ICU, complete ICU discharge CRF

   10. When patient is discharged from the hospital, complete Hospital discharge CRF.

   11. Day 60 and 90: Follow up about patient status. Complete phone follow-up CRF.

   Study population: Adult patients with COVID-19 diagnosed by PCR testing within previous 2 weeks and moderate to severe ARDS based on Berlin criteria (P/F < 200 while on PEEP ≥8 cm H2O) <48h in duration.

   Data Analysis: This is a pilot trial to determine whether patients with COVID-19-associated patients with ARDS should be included in a multicenter trial of TH+NMB in patients with ARDS from all causes. The data from this pilot will not be merged with data from the planned multicenter trial. The primary analysis of this pilot study will be to determine the effectiveness of the TH+NMB protocol in maintaining targeted temperature and to determine whether there are any safety issues with the TH+NMB protocol in this patient population.

   Data Management: Data for this pilot RCT will be recorded on paper CRFs. Completion of all fields will be checked in real-time. The forms have been designed to be compatible with the electronic versions developed for the multicenter trial.

   Randomization Plan: The investigators will use a randomization protocol stratified for proning status using pre-generated random assignment lists. Assignments will be made using an in-house Excel-based assignment tool, which blinds the observer to the assignment list.

   Subject Participation Duration: The duration of intervention, TH + NMB vs. usual temperature management, is 48h, followed by rewarming for 3-6h in the TH group. NMB will be discontinued and sedation reduced when subjects are rewarmed to core temperature ≥35.5°C. In the control group fever and hypothermia during continuous renal replacement therapy (CRRT) will be treated by protocol for 54h post-randomization. Physiologic and clinical parameters will be collected through study day 7. In hospital follow-up up to 90 days will include determination of 28-day VFDs and ICU-FDs, and day of hospital discharge. When the patient regains competence, consent for continued participation will be obtained

   Study Duration: Completion of enrollment is anticipated within 6 months.

ELIGIBILITY:
Inclusion Criteria for Enrollment

1. COVID-19 diagnosed by PCR within 3 weeks
2. men and women
3. any race/ethnicity
4. 18-65 years of age
5. endotracheal tube or tracheostomy in place and mechanically ventilated for < 7 days;
6. radiologic evidence of bilateral pulmonary infiltrates not fully explained by hydrostatic pulmonary edema
7. access to an LAR to provide consent (remote consent is permissible).

Additional inclusion criteria required for randomization:

1. meet all inclusion/exclusion criteria for enrollment
2. have a P/F ratio <200 with PEEP ≥8 cm H2O either from ABG or imputed from SpO2 as described by Brown et al (Chest 2016; 150:307).

Exclusion Criteria:

1. Missed ARDS window (>48hrs)
2. Missed mechanical ventilation window (>7 days)
3. Refractory hypotension (> 0.2 mcg/kg/min of norepinephrine or equivalent dose for minimum of 6 h)
4. Core temperature <35.5°C while not receiving CRRT
5. Patient is unable to give consent and no legally authorized representative is available;
6. Significant, active bleeding (>3u blood products and/or surgical/IR intervention)
7. Platelets <10K/mm3 (uncorrected)
8. Active hematologic malignancy
9. Skin process precludes cooling device
10. Moribund, not likely to survive 72h
11. Pre-morbid condition makes it unlikely that patient will survive 28 days
12. Do Not Resuscitate status
13. Not likely to remain intubated for ≥48h
14. Physician unwilling to participate
15. Severe underlying lung disease

    1. On home O2
    2. On BIPAP (except for OSA)
    3. Prior lung transplantation
16. BMI >45 kg/m2
17. Known NYHA class IV heart disease
18. Acute Coronary Syndrome past 30 days (MI, unstable angina)
19. Cardiac arrest within 30 days of enrollment
20. burns over >20% of the body surface
21. severe chronic liver disease (Child-Pugh of 12-15)
22. Previously randomized in CHILL study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-04-27 (Estimated); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Targeted temperature compliance | Randomization through day 3
  The total time in hours from beginning of cooling to beginning of rewarming during which the patient's core temperature was within the target range of 34-35°C.

SECONDARY OUTCOMES:
Adverse event | Randomization through study day 3
  Adverse events expected during cooling, including hemorrhage, bradycardia, and hypotension.
28-day ICU-free days | Calculated at study day 28 or death (whichever occurs first)
  Total number of days alive and not admitted to the ICU in the first 28 days after
Survival | calculated at 28, 60, and 90 days
  28-day, 60-day, and 90-day mortality
non neurologic Sequential Organ Failure (SOFA) scores | At enrollment and study days 1, 2, 3, 4, 7, and 28
  SOFA score excluding neurologic component - based on PaO2/FiO2 (0-4), BP and pressor requirement (0-4), bilirubin level (0-4), platelet count (0-4), and creatinine (0-14) with total composite score 0-20
Oxygen saturation (SpO2) | Measured at enrollment, every 4 hours on enrollment day, then once on day 2, 3, 4, 7 and 28
  Pulse ox reading
Plateau airway pressure | Measured at enrollment, every 4 hours on enrollment day, then once on day 2, 3, 4, and 7 or until extubation whichever occurs first
  On machine initiated breath
Mean airway pressure | Measured at enrollment, every 4 hours on enrollment day, then once on day 2, 3, 4, and 7 or until extubation whichever occurs first
  Direct ventilator measurement on machine initiated breath
Airway driving pressure | Measured at enrollment, every 4 hours on enrollment day, then once on day 2, 3, 4, and 7 or until extubation whichever occurs first
  Plateau pressure - PEEP (machine initiated breath)
Oxygen saturation index | Measured at enrollment, every 4 hours on enrollment day, then once on day 2, 3, 4, and 7 or until extubation whichever occurs first
  Mean airway pressure x 100 x FiO2/SpO2
Core temperature | Measured continuously and recorded at enrollment, every 2 hours on the day of enrollment, and mornings on study day 2, 3, 4, and 7
  Measured continuously from iv catheter, urinary catheter, or esophageal probe.
Urine output | Daily on study day 1, 2, 3, 4, and 7
  24 hour urine volume
comprehensive metabolic panel | Daily on study day 1, 2, 3, 4, and 7
  performed in clinical lab
Complete blood count with differential count and platelet count | Daily on study day 1, 2, 3, 4, and 7
  preformed in clinical lab
Biomarkers | Daily on study day 1, 2, 3, 4, and 7
  10 ml blood draw
Serum electrolytes | Every 8 hours until study hour 60
  performed in clinical lab
Blood glucose | Every 4 hours until study hour 60
  Beside blood glucose testing
28-day ventilator-free days | Calculated at study day 28 or death (whichever occurs first)
  Total number of days alive and not on a ventilator in the first 28 days after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D Hasday, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
At the completion of the study, Dr. Hasday and colleagues will present the results of the long-term outcomes at national meetings and publish them in peer-reviewed journals and in ClinicalTrials.gov. Within one year of the publication of the main trial data (whichever occurs first, Dr. Hasday will make de-identified study data available to any individual who presents an appropriate question and analysis plan. The available information will include 1) descriptive documents (e.g. study protocol, code book/variable dictionary, data collection instruments, and de-identification methodology), and 2) de-identified data file.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: All information will be available within one year of the publication of the main trial data.
Access Criteria: Access will either be by email to Dr. Hasday or through a website to be developed.

REFERENCES:
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Papazian L, Forel JM, Gacouin A, Penot-Ragon C, Perrin G, Loundou A, Jaber S, Arnal JM, Perez D, Seghboyan JM, Constantin JM, Courant P, Lefrant JY, Guerin C, Prat G, Morange S, Roch A; ACURASYS Study Investigators. Neuromuscular blockers in early acute respiratory distress syndrome. N Engl J Med. 2010 Sep 16;363(12):1107-16. doi: 10.1056/NEJMoa1005372. PMID 20843245
- [Background] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Background] Villar J, Blanco J, Kacmarek RM. Current incidence and outcome of the acute respiratory distress syndrome. Curr Opin Crit Care. 2016 Feb;22(1):1-6. doi: 10.1097/MCC.0000000000000266. PMID 26645551
- [Background] Hasday JD, Garrison A, Singh IS, Standiford T, Ellis GS, Rao S, He JR, Rice P, Frank M, Goldblum SE, Viscardi RM. Febrile-range hyperthermia augments pulmonary neutrophil recruitment and amplifies pulmonary oxygen toxicity. Am J Pathol. 2003 Jun;162(6):2005-17. doi: 10.1016/S0002-9440(10)64333-7. PMID 12759256
- [Background] Lipke AB, Matute-Bello G, Herrero R, Kurahashi K, Wong VA, Mongovin SM, Martin TR. Febrile-range hyperthermia augments lipopolysaccharide-induced lung injury by a mechanism of enhanced alveolar epithelial apoptosis. J Immunol. 2010 Apr 1;184(7):3801-13. doi: 10.4049/jimmunol.0903191. Epub 2010 Mar 3. PMID 20200273
- [Background] Lipke AB, Matute-Bello G, Herrero R, Wong VA, Mongovin SM, Martin TR. Death receptors mediate the adverse effects of febrile-range hyperthermia on the outcome of lipopolysaccharide-induced lung injury. Am J Physiol Lung Cell Mol Physiol. 2011 Jul;301(1):L60-70. doi: 10.1152/ajplung.00314.2010. Epub 2011 Apr 22. PMID 21515659
- [Background] Rice P, Martin E, He JR, Frank M, DeTolla L, Hester L, O'Neill T, Manka C, Benjamin I, Nagarsekar A, Singh I, Hasday JD. Febrile-range hyperthermia augments neutrophil accumulation and enhances lung injury in experimental gram-negative bacterial pneumonia. J Immunol. 2005 Mar 15;174(6):3676-85. doi: 10.4049/jimmunol.174.6.3676. PMID 15749906
- [Background] Shah NG, Tulapurkar ME, Damarla M, Singh IS, Goldblum SE, Shapiro P, Hasday JD. Febrile-range hyperthermia augments reversible TNF-alpha-induced hyperpermeability in human microvascular lung endothelial cells. Int J Hyperthermia. 2012;28(7):627-35. doi: 10.3109/02656736.2012.690547. Epub 2012 Jul 26. PMID 22834633
- [Background] Tulapurkar ME, Almutairy EA, Shah NG, He JR, Puche AC, Shapiro P, Singh IS, Hasday JD. Febrile-range hyperthermia modifies endothelial and neutrophilic functions to promote extravasation. Am J Respir Cell Mol Biol. 2012 Jun;46(6):807-14. doi: 10.1165/rcmb.2011-0378OC. Epub 2012 Jan 26. PMID 22281986
- [Background] Ball MK, Hillman NH, Kallapur SG, Polglase GR, Jobe AH, Pillow JJ. Body temperature effects on lung injury in ventilated preterm lambs. Resuscitation. 2010 Jun;81(6):749-54. doi: 10.1016/j.resuscitation.2009.12.007. Epub 2010 Mar 17. PMID 20299144
- [Background] Beurskens CJ, Aslami H, Kuipers MT, Horn J, Vroom MB, van Kuilenburg AB, Roelofs JJ, Schultz MJ, Juffermans NP. Induced hypothermia is protective in a rat model of pneumococcal pneumonia associated with increased adenosine triphosphate availability and turnover*. Crit Care Med. 2012 Mar;40(3):919-26. doi: 10.1097/CCM.0b013e3182373174. PMID 22036856
- [Background] Chang H, Huang KL, Li MH, Hsu CW, Tsai SH, Chu SJ. Manipulations of core temperatures in ischemia-reperfusion lung injury in rabbits. Pulm Pharmacol Ther. 2008;21(2):285-91. doi: 10.1016/j.pupt.2007.06.001. Epub 2007 Jun 14. PMID 17629529
- [Background] Chin JY, Koh Y, Kim MJ, Kim HS, Kim WS, Kim DS, Kim WD, Lim CM. The effects of hypothermia on endotoxin-primed lung. Anesth Analg. 2007 May;104(5):1171-8, tables of contents. doi: 10.1213/01.ane.0000260316.95836.1c. PMID 17456669
- [Background] Cruces P, Erranz B, Donoso A, Carvajal C, Salomon T, Torres MF, Diaz F. Mild hypothermia increases pulmonary anti-inflammatory response during protective mechanical ventilation in a piglet model of acute lung injury. Paediatr Anaesth. 2013 Nov;23(11):1069-77. doi: 10.1111/pan.12209. Epub 2013 Jun 3. PMID 23731357
- [Background] Huang PS, Tang GJ, Chen CH, Kou YR. Whole-body moderate hypothermia confers protection from wood smoke-induced acute lung injury in rats: the therapeutic window. Crit Care Med. 2006 Apr;34(4):1160-7. doi: 10.1097/01.CCM.0000207342.50559.0F. PMID 16484924
- [Background] Jo YH, Kim K, Rhee JE, Suh GJ, Kwon WY, Na SH, Alam HB. Therapeutic hypothermia attenuates acute lung injury in paraquat intoxication in rats. Resuscitation. 2011 Apr;82(4):487-91. doi: 10.1016/j.resuscitation.2010.11.028. Epub 2011 Jan 14. PMID 21236547
- [Background] Kim K, Kim W, Rhee JE, Jo YH, Lee JH, Kim KS, Kwon WY, Suh GJ, Lee CC, Singer AJ. Induced hypothermia attenuates the acute lung injury in hemorrhagic shock. J Trauma. 2010 Feb;68(2):373-81. doi: 10.1097/TA.0b013e3181a73eea. PMID 19996791
- [Background] Kira S, Daa T, Kashima K, Mori M, Noguchi T, Yokoyama S. Mild hypothermia reduces expression of intercellular adhesion molecule-1 (ICAM-1) and the accumulation of neutrophils after acid-induced lung injury in the rat. Acta Anaesthesiol Scand. 2005 Mar;49(3):351-9. doi: 10.1111/j.1399-6576.2005.00593.x. PMID 15752401
- [Background] Lim CM, Hong SB, Koh Y, Lee SD, Kim WS, Kim DS, Kim WD. Hypothermia attenuates vascular manifestations of ventilator-induced lung injury in rats. Lung. 2003;181(1):23-34. doi: 10.1007/s00408-002-0111-x. PMID 12879337
- [Background] Lim CM, Kim MS, Ahn JJ, Kim MJ, Kwon Y, Lee I, Koh Y, Kim DS, Kim WD. Hypothermia protects against endotoxin-induced acute lung injury in rats. Intensive Care Med. 2003 Mar;29(3):453-9. doi: 10.1007/s00134-002-1529-6. Epub 2002 Nov 22. PMID 12624664
- [Background] Peng CK, Huang KL, Wu CP, Li MH, Lin HI, Hsu CW, Tsai SH, Chu SJ. The role of mild hypothermia in air embolism-induced acute lung injury. Anesth Analg. 2010 May 1;110(5):1336-42. doi: 10.1213/ANE.0b013e3181d27e90. PMID 20418297
- [Background] Tang ZH, Hu JT, Lu ZC, Ji XF, Chen XF, Jiang LY, Zhang C, Jiang JS, Pang YP, Li CQ. Effect of mild hypothermia on the expression of toll-like receptor 2 in lung tissues with experimental acute lung injury. Heart Lung Circ. 2014 Dec;23(12):1202-7. doi: 10.1016/j.hlc.2014.05.016. Epub 2014 Jun 24. PMID 25224460
- [Background] Villar J, Slutsky AS. Effects of induced hypothermia in patients with septic adult respiratory distress syndrome. Resuscitation. 1993 Oct;26(2):183-92. doi: 10.1016/0300-9572(93)90178-s. PMID 8290813
- [Background] Karnatovskaia LV, Festic E, Freeman WD, Lee AS. Effect of therapeutic hypothermia on gas exchange and respiratory mechanics: a retrospective cohort study. Ther Hypothermia Temp Manag. 2014 Jun;4(2):88-95. doi: 10.1089/ther.2014.0004. Epub 2014 May 19. PMID 24840620
- [Background] Manthous CA, Hall JB, Olson D, Singh M, Chatila W, Pohlman A, Kushner R, Schmidt GA, Wood LD. Effect of cooling on oxygen consumption in febrile critically ill patients. Am J Respir Crit Care Med. 1995 Jan;151(1):10-4. doi: 10.1164/ajrccm.151.1.7812538.
- [Background] Gattinoni L, Tonetti T, Cressoni M, Cadringher P, Herrmann P, Moerer O, Protti A, Gotti M, Chiurazzi C, Carlesso E, Chiumello D, Quintel M. Ventilator-related causes of lung injury: the mechanical power. Intensive Care Med. 2016 Oct;42(10):1567-1575. doi: 10.1007/s00134-016-4505-2. Epub 2016 Sep 12. PMID 27620287
- [Background] Nagarsekar A, Tulapurkar ME, Singh IS, Atamas SP, Shah NG, Hasday JD. Hyperthermia promotes and prevents respiratory epithelial apoptosis through distinct mechanisms. Am J Respir Cell Mol Biol. 2012 Dec;47(6):824-33. doi: 10.1165/rcmb.2012-0105OC. Epub 2012 Sep 6. PMID 22962066
- [Background] Potla R, Singh IS, Atamas SP, Hasday JD. Shifts in temperature within the physiologic range modify strand-specific expression of select human microRNAs. RNA. 2015 Jul;21(7):1261-73. doi: 10.1261/rna.049122.114. Epub 2015 May 27. PMID 26018549
- [Background] Shah NG, Cowan MJ, Pickering E, Sareh H, Afshar M, Fox D, Marron J, Davis J, Herold K, Shanholtz CB, Hasday JD. Nonpharmacologic approach to minimizing shivering during surface cooling: a proof of principle study. J Crit Care. 2012 Dec;27(6):746.e1-8. doi: 10.1016/j.jcrc.2012.04.016. Epub 2012 Jul 2. PMID 22762936
- [Background] Beitler JR, Sands SA, Loring SH, Owens RL, Malhotra A, Spragg RG, Matthay MA, Thompson BT, Talmor D. Quantifying unintended exposure to high tidal volumes from breath stacking dyssynchrony in ARDS: the BREATHE criteria. Intensive Care Med. 2016 Sep;42(9):1427-36. doi: 10.1007/s00134-016-4423-3. Epub 2016 Jun 24. PMID 27342819
- [Background] Guerin C, Mancebo J. Prone positioning and neuromuscular blocking agents are part of standard care in severe ARDS patients: yes. Intensive Care Med. 2015 Dec;41(12):2195-7. doi: 10.1007/s00134-015-3918-7. Epub 2015 Sep 23. No abstract available. PMID 26399890
- [Background] Slack DF, Corwin DS, Shah NG, Shanholtz CB, Verceles AC, Netzer G, Jones KM, Brown CH, Terrin ML, Hasday JD. Pilot Feasibility Study of Therapeutic Hypothermia for Moderate to Severe Acute Respiratory Distress Syndrome. Crit Care Med. 2017 Jul;45(7):1152-1159. doi: 10.1097/CCM.0000000000002338. PMID 28406814
- [Background] Calfee CS, Ware LB, Eisner MD, Parsons PE, Thompson BT, Wickersham N, Matthay MA; NHLBI ARDS Network. Plasma receptor for advanced glycation end products and clinical outcomes in acute lung injury. Thorax. 2008 Dec;63(12):1083-9. doi: 10.1136/thx.2008.095588. Epub 2008 Jun 19. PMID 18566109
- [Background] Greene KE, Wright JR, Steinberg KP, Ruzinski JT, Caldwell E, Wong WB, Hull W, Whitsett JA, Akino T, Kuroki Y, Nagae H, Hudson LD, Martin TR. Serial changes in surfactant-associated proteins in lung and serum before and after onset of ARDS. Am J Respir Crit Care Med. 1999 Dec;160(6):1843-50. doi: 10.1164/ajrccm.160.6.9901117. PMID 10588595
- [Background] Calfee CS, Eisner MD, Parsons PE, Thompson BT, Conner ER Jr, Matthay MA, Ware LB; NHLBI Acute Respiratory Distress Syndrome Clinical Trials Network. Soluble intercellular adhesion molecule-1 and clinical outcomes in patients with acute lung injury. Intensive Care Med. 2009 Feb;35(2):248-57. doi: 10.1007/s00134-008-1235-0. Epub 2008 Aug 1. PMID 18670758
- [Background] Kimura D, Saravia J, Rovnaghi CR, Meduri GU, Schwingshackl A, Cormier SA, Anand KJ. Plasma Biomarker Analysis in Pediatric ARDS: Generating Future Framework from a Pilot Randomized Control Trial of Methylprednisolone: A Framework for Identifying Plasma Biomarkers Related to Clinical Outcomes in Pediatric ARDS. Front Pediatr. 2016 Mar 31;4:31. doi: 10.3389/fped.2016.00031. eCollection 2016. PMID 27066464
- [Background] Ferguson ND, Fan E, Camporota L, Antonelli M, Anzueto A, Beale R, Brochard L, Brower R, Esteban A, Gattinoni L, Rhodes A, Slutsky AS, Vincent JL, Rubenfeld GD, Thompson BT, Ranieri VM. The Berlin definition of ARDS: an expanded rationale, justification, and supplementary material. Intensive Care Med. 2012 Oct;38(10):1573-82. doi: 10.1007/s00134-012-2682-1. Epub 2012 Aug 25. PMID 22926653
- [Background] Brown SM, Grissom CK, Moss M, Rice TW, Schoenfeld D, Hou PC, Thompson BT, Brower RG; NIH/NHLBI PETAL Network Collaborators. Nonlinear Imputation of Pao2/Fio2 From Spo2/Fio2 Among Patients With Acute Respiratory Distress Syndrome. Chest. 2016 Aug;150(2):307-13. doi: 10.1016/j.chest.2016.01.003. Epub 2016 Jan 19. PMID 26836924

DOCUMENTS (3):
  • Study Protocol (2020-05-06): https://cdn.clinicaltrials.gov/large-docs/54/NCT03376854/Prot_013.pdf
  • Statistical Analysis Plan (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/54/NCT03376854/SAP_012.pdf
  • Informed Consent Form (2020-04-10): https://cdn.clinicaltrials.gov/large-docs/54/NCT03376854/ICF_011.pdf